CLINICAL TRIAL: NCT04653116
Title: Non-Interventional, Descriptive, Cross-sectional and Unicentric Study to Describe the Clinical Management in Asthmatic Patients Attended in the Influential Area of Hospital Universitario Virgen de la Victoria, Málaga
Brief Title: Clinical Management in Asthmatic Patients Attended in the Influential Area of Hospital Universitario Virgen de la Victoria, Málaga
Acronym: FIM-ASP-20201
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Other Study IDs: FIM-ASP-2020-01
Record Dates: First submitted 2020-11-20; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This evidence raises the need to determine the assistance quality care in asthma population in the influential area of Hospital Universitario Virgen de la Victoria through the assistance quality care indicators established by GEMA guidelines. The aim of this study is to obtain clinical data that allow to assess assistance quality degree in order to find improvement opportunities to achieve a better control of asthmatic patients within this influential area.

DETAILED DESCRIPTION:
Asthma is a heterogenic chronic disease characterized by acute symptomatic episodes of varying severity, including intermittently inflammation and narrowing of the airways in the lungs. The prevalence of this disease is high as affects more than 300 million people worldwide, which varies by country. In Spain, the prevalence it is estimated to be around 5%, ranged between 1% in Huelva and 4,7% in Albacete, according with the European Community Respiratory Survey (ECRHS), and seems to be increased due to a higher rate of asthma diagnosis1.

It's important to note that in this condition there is a substantial proportion of patients with inadequate control of their disease, which conducts to a higher morbidity and mortality2. The poor disease control is associated to an important negative impact in patient's health-related quality of life (HRQoL), causing them daily activity impairment, loss of work productivity and the need of using unscheduled doctor visits and hospital services3, 4. The direct and indirect costs in patients with a poor disease control represents an important proportion of the total cost of asthma, which it's estimated to be around 1-2% of the total public healthcare resources in developed countries, especially in patients with severe-persistent asthma4, 5.

The facts previously exposed turns this disease into a major public health problem due to its high prevalence within all age and sex groups and the high proportion of uncontrolled patients, which causes a high health burden to the National Health System, and which affects directly on the affected patients, as well as their families and the society6.

For this reason, during the past decades multiple clinical practice guidelines have been designed to improve the quality of care in patients with asthma and to reduce the high public burden associated to this disease7. International guidelines such as the Global Initiative for Asthma (GINA) and national guidelines as Guía Española para el Manejo del Asma (GEMA) in Spain, both of them stating that a good disease control can be achieved by most of asthma patients, were launched to increase the technical training of health professionals in order to reach a better disease management and conduct to a better quality of life in these patients 8, 9.

Specifically, GEMA guidelines also includes a tool to assess the level of assistance quality care through 8 indicators covering 4 dimensions: diagnose, non-pharmacological treatment, pharmacological treatment, monitoring.

However, since guidelines have been launched, there's still evidence of high proportion of patients with poorly disease control and large impact in patient's health-related quality of life10. Despite the availability of therapeutic recommendations through guidelines, clinical studies have shown that there's poor adherence to guidelines goals3. The Asthma Insight and Reality surveys, which were performed in several regions worldwide, concluded that all participating countries didn't met GINA goals. Specifically, in Central and Eastern Europe, the results showed a high proportion of asthma population who described physical activity limitations (68,2%) and acute symptoms during the previous 4 weeks (74%). Regarding disease monitoring, it' important to note that the results demonstrated that a 36,2% of asthmatic patients had never performed a lung function test11. A recent study conducted in Spain and Italy also evidenced a generally poor disease control, with around 50% of participant patients being considered uncontrolled12, and that strategies were needed to improve the management of this disease as it was concluded in a study performed in Spain to assess the disease control according to GINA criteria13.

In terms of costs, it's estimated that around 70% of the total cost of the disease is determined by this poor control and management14. An adequately disease management based in a higher use of preventive anti-inflammatory medication, a better education in asthma patients and an accurately follow of the recommendations of guidelines would result in a greater disease control and in a reduction of associated costs15, 16, 17.

This evidence raises the need to determine the assistance quality care in asthma population in the influential area of Hospital Universitario Virgen de la Victoria through the assistance quality care indicators established by GEMA guidelines. The aim of this study is to obtain clinical data that allow to assess assistance quality degree in order to find improvement opportunities to achieve a better control of asthmatic patients within this influential area.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with written informed consent prior to participation.
2. Patient female or male ≥ 18 years of age
3. Patient with asthma diagnosis more than one year before the study inclusion
4. Clinical data available at least 1 year before the study inclusion in the electronic medical records.

Exclusion Criteria:

1. Patient's participation in any clinical trial during the year prior to the index date for data collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed in Hospital Virgen de la Victoria, which it's the reference hospital that usually attends the asthma population of its influential area. Only patients that meet the eligibility criteria will be included in the study, and it is planned that a total estimation of 300 patients with asthma diagnose will be included in it. The whole patients will be recruited by the site investigator and collaborators, who will conduct the subject's medical chart review. Before the patient's study inclusion, the investigator team must have been obtained the signed informed consent (appendix 3) of each patient recruited and according to ICH GCP and to local legal requirements.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-29 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
To describe the clinical management in asthmatic | 6 month
  To describe the clinical management in asthmatic patients in the influential area of Hospital Universitario Virgen de la Victoria according to the assistant quality indicators established by GEMA guidelines

SECONDARY OUTCOMES:
To describe the sociodemographic and clinical characteristics | 6 month
  Age. Weight. Treatment. Exacerbations

CONTACTS AND LOCATIONS:
Locations (1):
- H. university virgen de la victoria, Málaga, Malaga, Spain